CLINICAL TRIAL: NCT03920904
Title: Peak Plasma Levels of Bupivacaine After a Pecto-Intercostal Fascial Block Post-Sternotomy for Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 19.015
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bupivacaine dosage in PIFB block: The pharmacokinetics of bupivacaine 0.25% with epinephrine 5 mcg/mL for a total dose of 2mg/kg of ideal body weight following a PIFB block will be determined by the collection of blood samples at predetermined time points.
  Interventions: Other: Collection of blood samples

INTERVENTIONS:
Other: Collection of blood samples — Nine blood samples will be collected to determine bupivacaine pharmacokinetics at T10min, T20min, T30min, T45min, T60min, T90min, T120min, T180min, and T240min. T0 will be defined as the end of bupivacaine injection.

SUMMARY:
The primary objective of the study is to measure plasma levels of bupivacaine following a pecto-intercostal fascial plane block (PIFB) in patients undergoing sternotomy for cardiac surgery.

DETAILED DESCRIPTION:
Heart disease such as ischemic cardiomyopathy and heart failure are the second leading cause of death and a leading cause of hospitalization in Canada. Approximately 35,000 heart valve or coronary artery revascularization procedures involving median sternotomy, an important component in the treatment of these diseases, are performed annually. Median sternotomy is associated with acute pain that decreases patient satisfaction, increases the risk of delirium, arrhythmias and respiratory complications. It also contributes to the development of postoperative chronic pain that can affect up to 31% of patients in the first year after surgery. Multimodal analgesia, combining drug therapy and regional anesthesia, can help in preventing acute and perhaps chronic pain in patients undergoing sternotomy for cardiac surgery.

The pecto-intercostal fascial plane block (PIFB) is a new locoregional anesthesia technique that has emerged to treat pain following cardiac surgery including sternotomy, breast surgeries and sternal fractures. It consists of injecting local anesthetics in the space located between the major pectoralis muscle and the intercostal muscles using ultrasound guidance, allowing to obtain anesthesia of the territory innervated by the anterior cutaneous intercostal branches, i.e. the medial aspect of the breast and the sternum.

The dose of local anesthetic injected after a PIFB should aim to maximize analgesia while minimizing the chance of toxic systemic concentrations. Defining the rate of absorption of local anesthetics into the blood after a PIFB will therefore help anesthesiologists to determinate optimal analgesic doses, in terms of both safety and effectiveness.

This observational study will determine bupivacaine pharmacokinetics after a PIFB with bupivacaine, to further define the right dose and duration of surveillance in post-anesthesia care.

Methods: Anesthesia and cardiac surgery will be initiated as usual. The use of bupivacaine by the anesthesiologist or surgeon will be prohibited. Following closure of the sternum, while the patient remains intubated and ventilated under general anesthesia with monitoring, including invasive blood pressure, oxygen saturation, respiratory rate and ECG, the PIFB will be done before application of sternal dressing and removal of sterile fields. Using an ultrasound machine with a high frequency linear probe (Sonosite, HFL50 15-6MHz) placed in the parasagittal plane, 3cm away from the midline, the fascia between the major pectoralis muscle and the internal intercostal muscle will be visualized. Subsequently, four injection sites, defined by the space between the fascia of the pectoral and intercostal muscles at the third and sixth intercostal spaces on each side of the patient, will be reached with an insulated hyperechoic needle (50-80 mm, 22 gauge, SonoPlex STIM, Nanoline, Pajunk, Germany) inserted cephalically and positioned in-plane.

Following negative aspiration, the anesthesiologist will confirm the correct position of the needle with the fluid spread of 1 mL of 5% dextrose. Then, he will inject bupivacaine 0.25% with epinephrine 5 mcg/mL in 5 ml aliquots for a total dose of 2mg/kg of ideal body weight (maximum of 150mg or 60 mL).

The end of injection will be considered as T0. Collection of 4.5mL of blood will be performed at T10min, T20min, T30min, T45min, T60min, T90min, T120min, T180min, and T240min.

Blood tubes will be immediately placed on ice to be ultimately sent to the laboratory for centrifugation and measurement of bupivacaine level using liquid chromatography-tandem mass spectrometry (LC-MS/MS) for each of the samples.

After the block, the patient will be transferred to the Intensive Care Unit. At T240min, if the patient is extubated, the level of the sensory block will be identified by the pinprick test.

The time between ICU arrival and extubation, as well as the total consumption of opioids and co-analgesics for the first 24 hours will be recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

* ASA l-lll
* Undergoing sternotomy for cardiac surgery under a PIFB and general anesthesia

Exclusion Criteria:

* Patient's refusal or inability to consent
* Allergy, hypersensibility or resistance to local anesthetic
* Contraindication to regional anesthesia: infection in the designated area, severe congenital coagulopathy or inadequate hemostasis before PIFB
* Severe hepatic (Child B and C) or renal insufficiency (GFR<30 mL/min)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a pecto-intercostal fascial block following cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Maximal plasma concentration (Cmax) of bupivacaine after pecto-intercostal fascial plane block | The end of injection of bupivacaine will be considered as T0. Blood samples at T10, T20, T30, T45, T60, T90, T120, T180, and T240minutes will be collected to further analyze plasmatic bupivacaine values at these timepoints.
  The Cmax will be estimated by interpolation based on the plasmatic bupivacaine values obtained after the analysis of the blood samples.

SECONDARY OUTCOMES:
Time (Tmax) to maximum plasma concentration Cmax of bupivacaine | The end of injection of bupivacaine will be considered as T0. Blood samples at T10, T20, T30, T45, T60, T90, T120, T180, and T240 minutes will be performed to further analyze plasmatic bupivacaine values at these timepoints.
  The Tmax will be estimated by interpolation based on the plasmatic bupivacaine values obtained after the analysis of the blood samples.
Total opioid and co-analgesics doses needed in the Intensive Care Unit | After the surgery, from the arrival in the Intensive Care Unit to 24 hours after the entry in the Intensive Care Unit.
  The total dose of opioids and co-analgesics used by the patients during the first 24 hours in the Intensive Care Unit will be recorded.
Time between arrival in Intensive Care Unit and extubation | Time from the arrival in the Intensive Care Unit to the extubation, for an average of 4 hours following surgery.
  Time between the arrival of the patient in the Intensive Care Unit and the extubation of the patient will be measured in minutes.
Sensory block level during the last sampling | At T240 minutes (4 hours) after the end of injection, after the last sampling, at the Intensive Care Unit
  Sensory block level will be measured with a 6.1g von Frey filaments.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Williams, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided